CLINICAL TRIAL: NCT01958775
Title: Regulation of Intestinal and Hepatic Lipoprotein Production by Glucagon Like
Brief Title: Regulation of Intestinal and Hepatic Lipoprotein Production by Glucagon Like Peptide 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: REB-07-0394
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Dyslipidemia
Keywords: Lipoproteins, apoB, GLP-2
MeSH Terms: conditions — Dyslipidemias | interventions — Glucagon-Like Peptide 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLP=2 (Experimental): active treatment with a single dose of GLP-2 (1500mcg)
  Interventions: Drug: GLP-2
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLP-2 — single subcutaneous dose of 1500mcg
  Other Names: glucagon like peptide 2
  Arms: GLP=2
Drug: Placebo
  Arms: Placebo

SUMMARY:
1. To assess whether Glucagon like peptide 2 (GLP-2) affects lipoprotein production (study A)
2. To assess whether GLP-2 affects the release of preformed chylomicrons (study B)

DETAILED DESCRIPTION:
Study A: Using constant feeding with a nasoduodenal tube and stable isotope infusion, mathematical modelling will be utilised to measure lipoprotein production and clearance. The lipoproteins assessed will be apoB-100 from the liver and apoB-48 from the intestine.

StudyB: Volunteers will be given a liquid meal with retinyl palmitate (vitamin A) to label chylomicrons made from the meal. 7 hours later they will be given GLP-2 or placebo. Measurements of plasma and TRL(triglyceride rich lipoprotein) triglyceride and TRL retinyl palmitate will be carried out to see whether GLP-2 increases these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Men and women, aged 18 to 60 years
  2. Body mass index 20 kg/m2 to 30 kg/m2
  3. Hemoglobin above 130g/L.
  4. Normal glucose tolerance in response to a 75g, 2-hr oral glucose tolerance test (OGTT)

Exclusion Criteria:

* 1. Subject has a history of hepatitis/hepatic disease that has been active within the previous two years.

  2. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL), genitourinary, hematological systems, or has severe uncontrolled treated or untreated hypertension (sitting diastolic BP > 100 or systolic > 180) or proliferative retinopathy 3. History of diabetes or OGTT indicative of diabetes or impaired glucose tolerance.

  4. Any history of ischemic heart disease or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or decompensated heart failure.

  5. Abnormal liver or thyroid function tests 6. Current addiction to alcohol or substances of abuse as determined by the investigator.

  7. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation 8. Taking any prescription or non-prescription medications at the time of the study 9. Having donated blood three months prior to and three months post study procedures 10. A pregnancy test will be performed 1 to 3 days prior to each study in all female research participants. Those who test positive for pregnancy will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Lipoprotein production and clearance rate | 10 hours
  ApoB 100 and ApoB 48 production and clearance

SECONDARY OUTCOMES:
Plasma and TRL triglyceride and TRL retinyl palmitate | 10 hours
  Measurements will be carried out hourly after ingestion of meal and then every 15-30 minutes thereafter to see if GLP-2 increases these parameters compared to placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dash S, Xiao C, Morgantini C, Connelly PW, Patterson BW, Lewis GF. Glucagon-like peptide-2 regulates release of chylomicrons from the intestine. Gastroenterology. 2014 Dec;147(6):1275-1284.e4. doi: 10.1053/j.gastro.2014.08.037. Epub 2014 Aug 28. PMID 25173752